CLINICAL TRIAL: NCT03744624
Title: Application of 3D Printing in Laparoscopic Surgery of Liver Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Jan Witowski, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122.6120.81.2017; 0054/DIA/2018/47 (Other Grant/Funding Number: Polish Ministry of Science and Higher Education)
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Liver Metastases
Keywords: 3D printing; Liver cancer; Laparoscopic surgery
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With 3D Model (Experimental): Patients in this arm will undergo laparoscopic liver resection with prior planning utilizing both 3D printed model and computed tomography (or/and magnetic resonance imaging)
  Interventions: Procedure: Laparoscopic liver resection; Device: 3D printing model
- Without 3D Model (Active Comparator): Patients in this arm will undergo laparoscopic liver resection with prior planning utilizing only standard medical imaging computed tomography (or/and magnetic resonance imaging) without development of 3D printed model
  Interventions: Procedure: Laparoscopic liver resection

INTERVENTIONS:
Procedure: Laparoscopic liver resection — Laparoscopic liver resection for oncological purposes
Device: 3D printing model — Use of 3D printed liver model in decision-making: preoperative planning and intraoperative guidance.
  Arms: With 3D Model

SUMMARY:
To explore the utility of personalized 3D printed liver models in planning and navigating laparoscopic resections.

DETAILED DESCRIPTION:
Project goal is to evaluate utility of personalized 3D printed models in preoperative planning and performing laparoscopic liver resections. Models will be developed with unique, low-cost approach. Project will consist of three overlapping modules/stages evaluating:

1. Accuracy of 3D printed liver models compared to computed tomography and standard surface or volume rendering
2. Whether 3D printed utilized in planning surgery affects the decision making regarding the surgical plan
3. Whether 3D printed models utilized in planning and navigating laparoscopic resections affect perioperative outcomes

Methodology of developing 3D models is described elsewhere. Printed models will be delivered to surgical team at least 5 days prior to the resection. Surgery will be performed in both arms according to the department's procedures and surgical oncology guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patient qualified to undergo liver tumor resection (either primary of metastatic; both benign and malignant lesions)
* Quality of imaging (CT or MRI or PET (positron emission tomography)/CT) satisfactory to develop 3D models
* Laparoscopic approach
* Informed consent

Exclusion Criteria:

* Open approach
* Technical limitations to model development
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of changes in surgery plan | intraoperative
Blood loss | intraoperative
Operative time | intraoperative

SECONDARY OUTCOMES:
Complications | intraoperative and until discharge, an average of 7 days
  Number of both total and severe (Clavien-Dindo>=3) complications
Length of stay | until patient discharge, an average of 7 days
Conversion rate | intraoperative
Readmissions | 6 months
Mortality | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of General Surgery Jagiellonian Univeristy Medical College, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Witowski JS, Pedziwiatr M, Major P, Budzynski A. Cost-effective, personalized, 3D-printed liver model for preoperative planning before laparoscopic liver hemihepatectomy for colorectal cancer metastases. Int J Comput Assist Radiol Surg. 2017 Dec;12(12):2047-2054. doi: 10.1007/s11548-017-1527-3. Epub 2017 Jan 31. PMID 28144830
- [Result] Witowski J, Wake N, Grochowska A, Sun Z, Budzynski A, Major P, Popiela TJ, Pedziwiatr M. Investigating accuracy of 3D printed liver models with computed tomography. Quant Imaging Med Surg. 2019 Jan;9(1):43-52. doi: 10.21037/qims.2018.09.16. PMID 30788245
- [Result] Witowski J, Budzynski A, Grochowska A, Ballard DH, Major P, Rubinkiewicz M, Zlahoda-Huzior A, Popiela TJ, Wierdak M, Pedziwiatr M. Decision-making based on 3D printed models in laparoscopic liver resections with intraoperative ultrasound: a prospective observational study. Eur Radiol. 2020 Mar;30(3):1306-1312. doi: 10.1007/s00330-019-06511-2. Epub 2019 Nov 26. PMID 31773294